CLINICAL TRIAL: NCT03706469
Title: A Phase 1, Open-Label, Randomized, Single Dose, 5-Period, 5-Treatment Study to Evaluate the Relative Bioavailability and Effect of Food on TAK-831 Tablet Formulations in Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability (BA) and Effect of Food on TAK-831 Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-831-1006; U1111-1217-5483 (Registry Identifier: WHO)
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fasted (T2 50 mg+T3 50 mg+T3 600 mg+T2 600 mg)+Fed (T3 600 mg) (Experimental): TAK-831 T2 50 milligram (mg), tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There will be a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
  Interventions: Drug: TAK-831 T2; Drug: TAK-831 T3
- Fasted (T3 50 mg+T2 600 mg+T2 50 mg+T3 600 mg)+Fed (T3 600 mg) (Experimental): TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There will be a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
  Interventions: Drug: TAK-831 T2; Drug: TAK-831 T3
- Fasted (T2 600 mg+T3 600 mg+T3 50 mg+T2 50 mg)+Fed (T3 600 mg) (Experimental): TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There will be a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
  Interventions: Drug: TAK-831 T2; Drug: TAK-831 T3
- Fasted (T3 600 mg+T2 50 mg+T2 600 mg+T3 50 mg)+Fed (T3 600 mg) (Experimental): TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There will be a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
  Interventions: Drug: TAK-831 T2; Drug: TAK-831 T3

INTERVENTIONS:
Drug: TAK-831 T2 — TAK-831 T2 Tablets.
Drug: TAK-831 T3 — TAK-831 T3 Tablets.

SUMMARY:
The purpose of this study is to assess the oral BA of TAK-831 T3 tablet formulation relative to TAK-831 T2 tablet formulation under fasting conditions and to assess the effect of food on the pharmacokinetics (PK) of TAK-831 T3 tablet formulation.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. TAK-831 is being tested in healthy participants to evaluate the relative BA and effect of food on the PK of TAK-831 tablet formulation.

The study will enroll approximately 16 participants. Participants will be randomly assigned (by chance, like flipping a coin) to TAK-831 in 1 of the 4 treatment sequences as following:

* T2 50 mg Fasted + T3 50 mg Fasted + T3 600 mg Fasted + T2 600 mg Fasted + T3 600 mg Fed
* T3 50 mg Fasted + T2 600 mg Fasted + T2 50 mg Fasted + T3 600 mg Fasted + T3 600 mg Fed
* T2 600 mg Fasted + T3 600 mg Fasted + T3 50 mg Fasted + T2 50 mg Fasted + T3 600 mg Fed
* T3 600 mg Fasted + T2 50 mg Fasted + T2 600 mg Fasted + T3 50 mg Fasted + T3 600 mg Fed

All participants will be asked to take tablet of assigned TAK-831 on Day 1 of each treatment period.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 70 days. Participants will make multiple visits to the clinic and will be contacted by clinic approximately 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than (<) 30.0 kilogram per square meter (kg/m^2), at Screening.

Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
2. Smokes more than 20 cigarettes or equivalent per day within 3 months prior to the first dose and is unwilling to discontinue use of any tobacco- or nicotine-containing products during the confinement period(s) of the study.
3. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
4. Is lactose intolerant or unable/unwilling to eat the high-fat breakfast.
5. Donation of blood or significant blood loss within 56 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 18 October 2018 to 22 December 2018.
Pre-assignment Details: Healthy participants were enrolled and randomized in one of the 4 treatment sequences to receive TAK-831.
Groups:
- Fasted (T2 50 mg+T3 50 mg+T3 600 mg+T2 600 mg)+Fed (T3 600 mg): TAK-831 T2 50 milligram (mg), tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There was a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
- Fasted (T3 50 mg+T2 600 mg+T2 50 mg+T3 600 mg)+Fed (T3 600 mg): TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There was a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
- Fasted (T2 600 mg+T3 600 mg+T3 50 mg+T2 50 mg)+Fed (T3 600 mg): TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There was a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
- Fasted (T3 600 mg+T2 50 mg+T2 600 mg+T3 50 mg)+Fed (T3 600 mg): TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There was a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
Period: Overall Study
Arm/Group | Fasted (T2 50 mg+T3 50 mg+T3 600 mg+T2 600 mg)+Fed (T3 600 mg) | Fasted (T3 50 mg+T2 600 mg+T2 50 mg+T3 600 mg)+Fed (T3 600 mg) | Fasted (T2 600 mg+T3 600 mg+T3 50 mg+T2 50 mg)+Fed (T3 600 mg) | Fasted (T3 600 mg+T2 50 mg+T2 600 mg+T3 50 mg)+Fed (T3 600 mg)
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of the study drug(s).
Groups:
- Fasted (T2 50 mg+T3 50 mg+T3 600 mg+T2 600 mg)+Fed (T3 600 mg): TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, followed by TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 2, followed by TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 3, followed by TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 4, further followed by TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5. There was a washout period of at least 7 days between study drug in-take in subsequent treatment periods.
- Total: Total of all reporting groups
Arm/Group | Fasted (T2 50 mg+T3 50 mg+T3 600 mg+T2 600 mg)+Fed (T3 600 mg) | Fasted (T3 50 mg+T2 600 mg+T2 50 mg+T3 600 mg)+Fed (T3 600 mg) | Fasted (T2 600 mg+T3 600 mg+T3 50 mg+T2 50 mg)+Fed (T3 600 mg) | Fasted (T3 600 mg+T2 50 mg+T2 600 mg+T3 50 mg)+Fed (T3 600 mg) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.94) | 49.0 (8.49) | 31.8 (9.22) | 30.0 (9.56) | 37.8 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 2 | 10
  Male | 3 | 0 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 3 | 4 | 4 | 4 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 16
Weight [Mean (Standard Deviation); unit: kilogram (Kg)] | 80.48 (9.694) | 67.55 (6.815) | 70.63 (19.643) | 76.07 (4.666) | 73.68 (11.660)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 175.3 (5.74) | 168.3 (6.65) | 169.5 (13.48) | 169.3 (2.06) | 170.6 (7.79)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.060 (1.6219) | 24.090 (4.1222) | 24.250 (3.3966) | 26.620 (1.9483) | 25.255 (2.8796)

OUTCOME MEASURES:

1. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hr/mL)
Groups:
- TAK-831 T2 50 mg Fasted: TAK-831 T2 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, 2, 3 or 4 as per assigned treatment sequence.
- TAK-831 T3 50 mg Fasted: TAK-831 T3 50 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, 2, 3 or 4 as per assigned treatment sequence.
- TAK-831 T2 600 mg Fasted: TAK-831 T2 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, 2, 3 or 4 as per assigned treatment sequence.
- TAK-831 T3 600 mg Fasted: TAK-831 T3 600 mg, tablet, orally, once, under fasted condition on Day 1 of Treatment Period 1, 2, 3 or 4 as per assigned treatment sequence.
- TAK-831 T3 600 mg Fed: TAK-831 T3 600 mg, tablet, orally, once, under fed condition on Day 1 of Treatment Period 5.
Arm/Group | TAK-831 T2 50 mg Fasted | TAK-831 T3 50 mg Fasted | TAK-831 T2 600 mg Fasted | TAK-831 T3 600 mg Fasted | TAK-831 T3 600 mg Fed
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nanogram*hour per milliliter(ng*hr/mL) | 714.8 (28.7) | 597.5 (37.0) | 4563 (24.8) | 4665 (41.8) | 8058 (29.0)
Statistical Analysis 1: Comparison: TAK-831 T2 50 mg Fasted vs TAK-831 T3 50 mg Fasted; Test type: Equivalence — Bioequivalence in the AUClast will be concluded if the 90 percent (%) confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; Percentage of Geometric Mean Ratio (GMR) = 83.60, 90% CI 2-sided [74.50 to 93.80]
Statistical Analysis 2: Comparison: TAK-831 T2 600 mg Fasted vs TAK-831 T3 600 mg Fasted; Test type: Equivalence — Bioequivalence in the AUClast will be concluded if the 90% confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; Percentage of GMR = 102.22, 90% CI 2-sided [91.10 to 114.70]
Statistical Analysis 3: Comparison: TAK-831 T3 600 mg Fasted vs TAK-831 T3 600 mg Fed; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage of GMR = 172.73, 90% CI 2-sided [152.55 to 195.58]

2. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration. The PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-831 T2 50 mg Fasted | TAK-831 T3 50 mg Fasted | TAK-831 T2 600 mg Fasted | TAK-831 T3 600 mg Fasted | TAK-831 T3 600 mg Fed
Number analyzed (Participants) | 14 | 11 | 16 | 14 | 15
ng*hr/mL | 761.8 (29.3) | 688.6 (31.0) | 4665 (26.0) | 4558 (41.8) | 7934 (27.3)
Statistical Analysis 1: Comparison: TAK-831 T2 50 mg Fasted vs TAK-831 T3 50 mg Fasted; Test type: Equivalence — Bioequivalence in the AUC∞ will be concluded if the 90% confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; Percentage of GMR = 84.29, 90% CI 2-sided [73.92 to 96.11]
Statistical Analysis 2: Comparison: TAK-831 T2 600 mg Fasted vs TAK-831 T3 600 mg Fasted; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Percentage of GMR = 99.61, 90% CI 2-sided [88.88 to 111.63]
Statistical Analysis 3: Comparison: TAK-831 T3 600 mg Fasted vs TAK-831 T3 600 mg Fed; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Percentage of GMR = 172.70, 90% CI 2-sided [149.07 to 200.09]

3. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK analysis set included all participants from the safety set who had at least 1 measurable postdose TAK-831 plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-831 T2 50 mg Fasted | TAK-831 T3 50 mg Fasted | TAK-831 T2 600 mg Fasted | TAK-831 T3 600 mg Fasted | TAK-831 T3 600 mg Fed
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nanogram per milliliter (ng/mL) | 397.5 (38.8) | 314.6 (40.0) | 1384 (28.9) | 1381 (24.6) | 2394 (37.1)
Statistical Analysis 1: Comparison: TAK-831 T2 50 mg Fasted vs TAK-831 T3 50 mg Fasted; Test type: Equivalence — Bioequivalence in the Cmax will be concluded if the 90% confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; Percentage of GMR = 79.14, 90% CI 2-sided [67.36 to 92.99]
Statistical Analysis 2: Comparison: TAK-831 T2 600 mg Fasted vs TAK-831 T3 600 mg Fasted; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Percentage of GMR = 99.80, 90% CI 2-sided [84.94 to 117.27]
Statistical Analysis 3: Comparison: TAK-831 T3 600 mg Fasted vs TAK-831 T3 600 mg Fed; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Percentage of GMR = 173.30, 90% CI 2-sided [150.05 to 200.16]

4. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Day 1 post dose up to 14 days after the last dose of study drug (Up to Day 47)
Population: The safety analysis set included all participants who received at least one dose of the study drug(s).
Measure: Number; unit: percentage of participants
Arm/Group | TAK-831 T2 50 mg Fasted | TAK-831 T3 50 mg Fasted | TAK-831 T2 600 mg Fasted | TAK-831 T3 600 mg Fasted | TAK-831 T3 600 mg Fed
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
percentage of participants | 0 | 13 | 0 | 6 | 0

ADVERSE EVENTS:
Time Frame: Day 1 post dose up to 14 days after the last dose of study drug ( Up to Day 47).
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report adverse events occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-831 T2 50 mg Fasted | TAK-831 T3 50 mg Fasted | TAK-831 T2 600 mg Fasted | TAK-831 T3 600 mg Fasted | TAK-831 T3 600 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16 | 0/16 | 1/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-831 T2 50 mg Fasted (N=16) | TAK-831 T3 50 mg Fasted (N=16) | TAK-831 T2 600 mg Fasted (N=16) | TAK-831 T3 600 mg Fasted (N=16) | TAK-831 T3 600 mg Fed (N=16)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03706469/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03706469/SAP_001.pdf